CLINICAL TRIAL: NCT03109171
Title: Accuracy of the Sensory Test Performed Using the Laryngopharyngeal Endoscopic Esthesiometer and Rangefinder in Patients With Suspected Obstructive Sleep Apnoea Hypopnea (OSA): a Prospective Double-blinded, Randomised, Pilot Study
Brief Title: Accuracy of the Sensory Test Using the Laryngopharyngeal Endoscopic Esthesiometer in Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Neumologica Colombiana (Other)
Collaborators: Universidad de la Sabana (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, Luis F. Giraldo-Cadavid, Pulmonologist, Fundación Neumologica Colombiana
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 201611-22405
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sleep Apnea, Obstructive; Larynx; Sensory Disorder
Keywords: Endoscopy; Lasers; Fiber Optic Technology; Bronchoscopy; Esthesiometer; Mechanoreceptors; Diagnosis; Reflex; Reproducibility of Results; Reliability of Results; Validity of Results; Sensory Thresholds
MeSH Terms: conditions — Sleep Apnea, Obstructive; Laryngeal Diseases; Sensation Disorders; Disease

STUDY DESIGN:
Intervention Model Description: Subjects participating in the inter-rater reliability evaluation will be evaluated by two raters, an expert and a non-expert rater, each rater performing two measurements of laryngopharyngeal sensory thresholds (ST) two times at each side (right and left) of the corresponding laryngopharyngeal structure. All other subjects, participating in the accuracy evaluation, will be evaluated by only one expert rater who will perform three measurements of laryngopharyngeal ST per subject. The varying degrees of rater experience aims to reproduce common scenarios when a new technique (like the measurement of laryngopharyngeal mechanosensitivity) is introduced to clinical practice.
  The two raters will measure the ST sequentially and in a randomized cross-over design in each subject (the order in which each rater intervenes will be randomized) aiming that the sensory tests be started an equal number of times by an expert rater and non-expert rater.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation sequence, determining which rater (expert vs non-expert) intervenes first or second, will be concealed using the SNOSE strategy (sequentially numbered opaque sealed envelopes). One of the authors (ARB), who has not competing interests will generate the allocation sequence and conceal it in envelopes. While the first rater measures the sensory thresholds (ST) the second rater will be at a different room for blinding purposes. There will be no communication about the testing results between the two raters nor the staff who are helping the testing performance.
  To mask the values of the ST, air pulses will be identified by a random combination of three letters instead of by the intensity levels corresponding to the air pulses. The raters will not know the intensity corresponding to each letter combination. At the end of the test, an assistant will replace the letters corresponding to the ST values by the intensity levels of the air pulses in units of force (millinewtons)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expert rater (Other): Pulmonologist or Otolaryngologist with experience in laryngopharyngeal sensory evaluation: who has made more than 50 laryngopharyngeal sensory tests.
  Interventions: Other: Laryngopharyngeal sensory test
- Non-expert rater (Other): * Pulmonologist or Otolaryngologist inexperienced in laryngopharyngeal sensory evaluation: who has made minimum 5 and maximum 50 laryngopharyngeal sensory tests.
  * Pulmonologist fellow who has completed the training provided for a Pulmonologist Fellow in bronchoscopy and who has performed minimum 5 and maximum 50 laryngopharyngeal sensory testing.
  Interventions: Other: Laryngopharyngeal sensory test

INTERVENTIONS:
Other: Laryngopharyngeal sensory test — The sensory measurements will include thresholds for psychophysical sensory thresholds at the velopharynx, hypopharynx and aryepiglottic folds

SUMMARY:
This is a prospective double blinded randomized crossover controlled trial aiming at validating the measurement of laryngopharyngeal mechanosensitivity in patients with suspected OSA using a recently developed laryngopharyngeal endoscopic esthesiometer and rangefinder (LPEER).

Subjects will be recruited from patients with suspected OSA referred for baseline polysomnography to a university hospital sleep laboratory. Intra- and inter-rater reliability will be evaluated using the Bland-Altman's limits of agreement plot, the intraclass correlation coefficient, and the Pearson or Spearman correlation coefficient, depending on the distribution of the variables. Diagnostic accuracy will be evaluate plotting Receiver-operating-characteristic-curves (ROC-curves) using as reference standard basal polysomnogram. The sensory threshold values for patients with mild, moderate, and severe OSA, will be determined and compared using ANOVA or Kruskal Wallis test, depending on the distribution of the variables.

DETAILED DESCRIPTION:
INTRODUCTION:

Obstructive sleep apnea-hypopnea syndrome (OSA) patients might have varying degrees of laryngopharyngeal mechanical hyposensitivity; however, these findings come from studies performed with methods having weak inter-rater reliability and accuracy evidence.

The purpose of this study is to validate the measurement of laryngopharyngeal mechanosensitivity in patients with OSA using a recently developed laryngopharyngeal endoscopic esthesiometer and rangefinder (LPEER). The LPEER includes an air-pulse generator and an endoscopic laser rangefinder and works coupled to a conventional fiberoptic endoscope. This device generates air-pulses ranging from 0.04 mN to 16.5 mN in order to cover a wide range of laryngopharyngeal reflexes and sensory thresholds. Depending on the reflex or sensory threshold to be explored the LPEER is configured to deliver a sequence of 10 air-pulses of different intensity.

METHODS:

The study will be prospective, double blinded, and with a randomized and crossover assignment of the raters.

Subjects will be recruited from patients with suspected OSA referred for baseline polysomnography to a sleep laboratory of a tertiary care university hospital. They will undergo a laryngopharyngeal sensory test using the LPEER, which includes measurement of the thresholds for the velopharyngeal, hypopharyngeal and aryepiglottic fold psychophysical sensitivity.

Intra- and inter-rater reliability will be evaluated using the Bland-Altman's limits of agreement plot, the intraclass correlation coefficient, and the Pearson or Spearman correlation coefficient, depending on the distribution of the variables.

Diagnostic accuracy will be evaluate plotting ROC-curves using as reference standard basal polysomnogram. The sensory threshold values for patients with mild, moderate, and severe OSA, will be determined and compared using ANOVA or Kruskal Wallis test, depending on the distribution of the variables.The discriminative capacity as well as correlations between laryngopharyngeal sensory thresholds and OSA severity indexes will be explored in subgroups of subjects with normal and abnormal sensation. The relationship between sensory thresholds and OSA severity indexes will be explored by linear equations as well as by second- and higher-order polynomial equations.

The laryngopharyngeal endoscopic esthesiometer and rangefinder (LPEER), could be a new tool for the evaluation and monitoring of laryngopharyngeal sensory involvement in patients with OSA, which, if proved valid, could help to increase the knowledge about the pathophysiological mechanisms of this condition and potentially help finding new therapeutic interventions for OSA.

ETHICS:

This study will follow the Declaration of Helsinki principles and national legal regulations about research in human subjects. The protocol was approved by the Institutional Review Board of Fundacion Neumologica Colombiana and all recruited subjects will provided a signed informed consent.

DISSEMINATION:

The results will be disseminated through conference presentations and peer-reviewed publication.

ELIGIBILITY:
Inclusion Criteria:

* Patients being 18 years old or more referred to the sleep laboratory of a tertiary care university hospital for a baseline polysomnography for suspected OSA.

Exclusion Criteria:

* Anticoagulation (though not a contraindication for the endoscopic laryngopharyngeal sensory test, anticoagulation is an exclusion criteria for this validation study in order to keep it a minimal-risk study).
* Bleeding diathesis.
* Basal awake oxygen saturation by pulse oximetry below 88%.
* Not agree to participate in the study.
* Glasgow coma scale below of 15 (to avoid confusion with involvement of laryngopharyngeal reflexes due to neurological disease accompanied by decreased level of consciousness).
* Baseline polysomnography that does not meet validity criteria to be interpreted (according to the American Academy of Sleep Medicine).
* Baseline polysomnography performed more than 15 days before the sensory testing. Ordinarily, the sensory testing will be performed the same day or the next day of baseline polysomnography.
* More than 5% of total apnoea events being of central origin.
* History of maxillofacial or pharyngeal surgery (to avoid confusion with involvement of laryngopharyngeal reflexes due to surgery in this region).
* Laryngopharyngeal tract malignancies (to avoid confusion with involvement of laryngopharyngeal reflexes due to tumours).
* Central Nervous System (CNS) surgery in the last three months or that has left neurological sequelae (to avoid confusion with involvement of laryngopharyngeal reflexes due to sequelae of CNS surgery).
* Traumatic brain injury in the last three months or more than three month with neurological sequelae.
* History of active neuromuscular disease that affects the muscles of head and neck or with sequels present at the time of the sensory testing (to avoid confusion with involvement of laryngopharyngeal reflexes due to neuromuscular disease).
* History of cerebrovascular disease (to avoid confusion with dysphagia or sensory compromise secondary to cerebrovascular disease).
* Diabetes (to avoid confusion with diabetic neuropathy that compromises the laryngopharyngeal region).
* Chronic use of systemic corticosteroids at a dose greater or equal to 20 mg per day of prednisone or equivalent (to avoid confusion with steroid myopathy that compromises the laryngopharyngeal region).
* Upper respiratory tract infection within 15 days prior to the testing (to avoid confusion with neuropathy associated with respiratory viral disease that compromises the laryngopharyngeal region).
* Patient's inability to cooperate during the examination (to avoid measurement error caused by the lack of cooperation of the patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Velopharynx psychophysical sensory threshold | 15 days
  Sensitivity threshold at the velopharynx in millinewtons (mN).
Hypopharynx psychophysical sensory threshold | 15 days
  Sensitivity threshold at the hypopharynx in millinewtons (mN).
Aryepiglottic fold psychophysical sensory threshold | 15 days
  Sensitivity threshold at the aryepiglottic folds in millinewtons (mN).

SECONDARY OUTCOMES:
Apnea Hypopnea Index | 15 days
  Number of apneas and hypopneas per hour reported in polysomnography, according to the American Academy of Sleep Medicine criteria.
Oxygen desaturation index | 15 days
  Number of desaturation episodes by pulse oximetry (SpO2%) (>3% fall in SpO2%) per hour reported in polysomnography, according to the American Academy of Sleep Medicine criteria.
T90 | 15 days
  Time spent at oxygen saturation below 90% by pulse oximetry
Adverse Events | 15 days
  Any adverse event potentially related to the laryngopharyngeal sensory test, including pain, gagging, discomfort, laryngospasm, syncope or pre-syncope, epistaxis, need for observation or referral to emergency room or hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Giraldo-Cadavid, MD, PhD, Study Chair — University of La Sabana; Fundacion Neumologica Colombiana
Locations (2):
- Colombia (2):
  - Fundacion Neumologica Colombiana, Bogotá, Bogota D.C.
  - Universidad de la Sabana, Chía, Cundinamarca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miyaji H, Hironaga N, Umezaki T, Hagiwara K, Shigeto H, Sawatsubashi M, Tobimatsu S, Komune S. Neuromagnetic detection of the laryngeal area: Sensory-evoked fields to air-puff stimulation. Neuroimage. 2014 Mar;88:162-9. doi: 10.1016/j.neuroimage.2013.11.008. Epub 2013 Nov 15. PMID 24246493
- [Background] Nguyen AT, Jobin V, Payne R, Beauregard J, Naor N, Kimoff RJ. Laryngeal and velopharyngeal sensory impairment in obstructive sleep apnea. Sleep. 2005 May;28(5):585-93. doi: 10.1093/sleep/28.5.585. PMID 16171271
- [Background] Aviv JE, Martin JH, Sacco RL, Zagar D, Diamond B, Keen MS, Blitzer A. Supraglottic and pharyngeal sensory abnormalities in stroke patients with dysphagia. Ann Otol Rhinol Laryngol. 1996 Feb;105(2):92-7. doi: 10.1177/000348949610500202. PMID 8659942
- [Background] Aviv JE, Sacco RL, Mohr JP, Thompson JL, Levin B, Sunshine S, Thomson J, Close LG. Laryngopharyngeal sensory testing with modified barium swallow as predictors of aspiration pneumonia after stroke. Laryngoscope. 1997 Sep;107(9):1254-60. doi: 10.1097/00005537-199709000-00018. PMID 9292613
- [Background] Jordan AS, McSharry DG, Malhotra A. Adult obstructive sleep apnoea. Lancet. 2014 Feb 22;383(9918):736-47. doi: 10.1016/S0140-6736(13)60734-5. Epub 2013 Aug 2. PMID 23910433
- [Background] Teramoto S, Sudo E, Matsuse T, Ohga E, Ishii T, Ouchi Y, Fukuchi Y. Impaired swallowing reflex in patients with obstructive sleep apnea syndrome. Chest. 1999 Jul;116(1):17-21. doi: 10.1378/chest.116.1.17. PMID 10424498
- [Background] Valbuza JS, de Oliveira MM, Zancanella E, Conti CF, Prado LB, Carvalho LB, do Prado GF. Swallowing dysfunction related to obstructive sleep apnea: a nasal fibroscopy pilot study. Sleep Breath. 2011 May;15(2):209-13. doi: 10.1007/s11325-010-0474-9. Epub 2011 Jan 13. PMID 21229321
- [Background] Giraldo-Cadavid LF, Burguete J, Rueda F, Galvis AM, Castaneda N, Agudelo-Otalora LM, Moscoso WD, Paez N, Fernandez S. Reliability of a laryngo-pharyngeal esthesiometer and a method for measuring laryngo-pharyngeal mechano-sensitivity in a prospectively recruited cohort of patients. Eur Arch Otorhinolaryngol. 2017 Jul;274(7):2861-2870. doi: 10.1007/s00405-017-4536-5. Epub 2017 Mar 24. PMID 28341965
- [Background] Giraldo-Cadavid LF, Agudelo-Otalora LM, Burguete J, Arbulu M, Moscoso WD, Martinez F, Ortiz AF, Diaz J, Pantoja JA, Rueda-Arango AF, Fernandez S. Design, development and validation of a new laryngo-pharyngeal endoscopic esthesiometer and range-finder based on the assessment of air-pulse variability determinants. Biomed Eng Online. 2016 May 10;15(1):52. doi: 10.1186/s12938-016-0166-1. PMID 27160751
- [Background] Oliveira LA, Fontes LH, Cahali MB. Swallowing and pharyngo-esophageal manometry in obstructive sleep apnea. Braz J Otorhinolaryngol. 2015 May-Jun;81(3):294-300. doi: 10.1016/j.bjorl.2015.03.006. Epub 2015 Mar 30. PMID 25921934
- [Background] Chien MY, Wu YT, Lee PL, Chang YJ, Yang PC. Inspiratory muscle dysfunction in patients with severe obstructive sleep apnoea. Eur Respir J. 2010 Feb;35(2):373-80. doi: 10.1183/09031936.00190208. Epub 2009 Jul 30. PMID 19643936
- [Background] Tsai YJ, Ramar K, Liang YJ, Chiu PH, Powell N, Chi CY, Lung TC, Wen-Yang Lin W, Tseng PJ, Wu MY, Chien KC, Weaver EM, Lee FP, Lin CM, Chen KC, Chiang RP. Peripheral neuropathology of the upper airway in obstructive sleep apnea syndrome. Sleep Med Rev. 2013 Apr;17(2):161-8. doi: 10.1016/j.smrv.2012.05.005. Epub 2012 Aug 17. PMID 22902356
- [Background] Eckert DJ, Lo YL, Saboisky JP, Jordan AS, White DP, Malhotra A. Sensorimotor function of the upper-airway muscles and respiratory sensory processing in untreated obstructive sleep apnea. J Appl Physiol (1985). 2011 Dec;111(6):1644-53. doi: 10.1152/japplphysiol.00653.2011. Epub 2011 Sep 1. PMID 21885797
- [Background] Fogel RB, Malhotra A, Shea SA, Edwards JK, White DP. Reduced genioglossal activity with upper airway anesthesia in awake patients with OSA. J Appl Physiol (1985). 2000 Apr;88(4):1346-54. doi: 10.1152/jappl.2000.88.4.1346. PMID 10749829
- [Background] Kezirian EJ, Boudewyns A, Eisele DW, Schwartz AR, Smith PL, Van de Heyning PH, De Backer WA. Electrical stimulation of the hypoglossal nerve in the treatment of obstructive sleep apnea. Sleep Med Rev. 2010 Oct;14(5):299-305. doi: 10.1016/j.smrv.2009.10.009. Epub 2010 Jan 29. PMID 20116305
- [Background] Gillick BT, Zirpel L. Neuroplasticity: an appreciation from synapse to system. Arch Phys Med Rehabil. 2012 Oct;93(10):1846-55. doi: 10.1016/j.apmr.2012.04.026. Epub 2012 May 18. PMID 22613094
- [Background] Page SJ, Cunningham DA, Plow E, Blazak B. It takes two: noninvasive brain stimulation combined with neurorehabilitation. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S89-93. doi: 10.1016/j.apmr.2014.09.019. PMID 25813373
- [Background] Robbins SM, Houghton PE, Woodbury MG, Brown JL. The therapeutic effect of functional and transcutaneous electric stimulation on improving gait speed in stroke patients: a meta-analysis. Arch Phys Med Rehabil. 2006 Jun;87(6):853-9. doi: 10.1016/j.apmr.2006.02.026. PMID 16731222
- [Background] Howlett OA, Lannin NA, Ada L, McKinstry C. Functional electrical stimulation improves activity after stroke: a systematic review with meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):934-43. doi: 10.1016/j.apmr.2015.01.013. Epub 2015 Jan 26. PMID 25634620
- [Background] Gallas S, Marie JP, Leroi AM, Verin E. Sensory transcutaneous electrical stimulation improves post-stroke dysphagic patients. Dysphagia. 2010 Dec;25(4):291-7. doi: 10.1007/s00455-009-9259-3. Epub 2009 Oct 24. PMID 19856025
- [Background] Rofes L, Arreola V, Lopez I, Martin A, Sebastian M, Ciurana A, Clave P. Effect of surface sensory and motor electrical stimulation on chronic poststroke oropharyngeal dysfunction. Neurogastroenterol Motil. 2013 Nov;25(11):888-e701. doi: 10.1111/nmo.12211. Epub 2013 Aug 12. PMID 23937476
- [Background] Aviv JE, Martin JH, Keen MS, Debell M, Blitzer A. Air pulse quantification of supraglottic and pharyngeal sensation: a new technique. Ann Otol Rhinol Laryngol. 1993 Oct;102(10):777-80. doi: 10.1177/000348949310201007. PMID 8215097
- [Background] Cunningham JJ, Halum SL, Butler SG, Postma GN. Intraobserver and interobserver reliability in laryngopharyngeal sensory discrimination thresholds: a pilot study. Ann Otol Rhinol Laryngol. 2007 Aug;116(8):582-8. doi: 10.1177/000348940711600805. PMID 17847725
- [Background] Hammer MJ. Design of a new somatosensory stimulus delivery device for measuring laryngeal mechanosensory detection thresholds in humans. IEEE Trans Biomed Eng. 2009 Apr;56(4):1154-9. doi: 10.1109/TBME.2008.2007968. Epub 2008 Oct 31. PMID 19272888
- [Background] Larsson H, Carlsson-Nordlander B, Lindblad LE, Norbeck O, Svanborg E. Temperature thresholds in the oropharynx of patients with obstructive sleep apnea syndrome. Am Rev Respir Dis. 1992 Nov;146(5 Pt 1):1246-9. doi: 10.1164/ajrccm/146.5_Pt_1.1246. PMID 1443879
- [Background] Kimoff RJ, Sforza E, Champagne V, Ofiara L, Gendron D. Upper airway sensation in snoring and obstructive sleep apnea. Am J Respir Crit Care Med. 2001 Jul 15;164(2):250-5. doi: 10.1164/ajrccm.164.2.2010012. PMID 11463596
- [Background] Aviv JE, Murry T, Zschommler A, Cohen M, Gartner C. Flexible endoscopic evaluation of swallowing with sensory testing: patient characteristics and analysis of safety in 1,340 consecutive examinations. Ann Otol Rhinol Laryngol. 2005 Mar;114(3):173-6. doi: 10.1177/000348940511400301. PMID 15825564
- [Derived] Giraldo-Cadavid LF, Bastidas AR, Padilla-Ortiz DM, Concha-Galan DC, Bazurto MA, Vargas L. Accuracy and reliability of the sensory test performed using the laryngopharyngeal endoscopic esthesiometer and rangefinder in patients with suspected obstructive sleep apnoea hypopnoea: protocol for a prospective double-blinded, randomised, exploratory study. BMJ Open. 2017 Aug 21;7(8):e015235. doi: 10.1136/bmjopen-2016-015235. PMID 28827237
- See also: Endoscopic Laryngopharyngeal Sensory Test (ELST) Protocol for the Validation of a Laryngo-Pharyngeal Endoscopic Esthesiometer and Rangefinder (LPEER) — https://upperairwaylfgiraldo.wordpress.com/about/